CLINICAL TRIAL: NCT02632552
Title: A Technology-Assisted Care Transition Intervention for Veterans With Chronic Heart Failure or Chronic Obstructive Pulmonary Disease
Brief Title: A Technology Assisted Care Transition Intervention for Veterans With CHF or COPD
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-101
Record Dates: First submitted 2015-12-11; First posted 2015-12-16 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: CHF; COPD
Keywords: care transition; technology; chronic heart failure; chronic obstructive pulmonary disease; virtual nurse; texting; informatics; Veterans
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Technology-assisted care transition arm (Experimental): In-patient virtual nurse on-screen touchscreen and outpatient virtual nurse follow-up by texting
  Interventions: Behavioral: Technology-assisted care transition intervention
- Active attention control (Active Comparator): In-patient brief animated power-point style didactic onscreen tutorial covering the core pillars of care transitions and brief outpatient texting
  Interventions: Behavioral: Active attention control

INTERVENTIONS:
Behavioral: Technology-assisted care transition intervention — In-patient virtual nurse on-screen touchscreen and outpatient virtual nurse follow-up by texting
  Other Names: Virtual Nurse Annie Fox Intervention
  Arms: Technology-assisted care transition arm
Behavioral: Active attention control — In-patient brief animated power-point style didactic onscreen tutorial covering the core pillars of care transitions and brief outpatient texting
  Arms: Active attention control

SUMMARY:
Transition from hospital to home places patients in jeopardy of adverse events and increases their risk for rehospitalization. CHF is the most prevalent chronic condition among U.S. adults and COPD is the third leading cause of death in the U.S. Both CHF and COPD represent significant burdens for the VHA healthcare system. Care transitions can be supported through multi-component interventions, but are costly to implement. Virtual nurses provide an effective medium for explaining health concepts to patients, and previous work indicates patients find virtual nurses acceptable. The investigators will implement and evaluate a virtual nurse intervention to provide automated, tailored, and timely support to Veterans transitioning from hospital to home. As effective care transition interventions incorporate both inpatient and outpatient components, the virtual nurse will first engage with patient onscreen during their inpatient stay and then via text message post-discharge. This project has the potential to improve the care transition experience for patients, caregivers and healthcare providers.

DETAILED DESCRIPTION:
The last decade has seen a steady increase in the resources that VHA uses to treat chronic heart failure (CHF) and Chronic Obstructive Pulmonary Disease (COPD), both of which are among the most common reasons for admission and re-admission in VHA facilities. Multi-component care transition interventions can be effective, but are costly. One approach to reduce complexity and costs is to offload some work to technology.

Informed by the sociotechnical model, this study proposes a technology-assisted care transition intervention founded on the concept of a virtual nurse that interacts with Veterans through different technology channels. The virtual nurse is an anthropomorphized computer program designed to simulate a discharge nurse. During the inpatient stay, the virtual nurse will appear on a computer touch screen and will educate Veterans with CHF or COPD about the important components of a care transition (drawing on the Coleman Care Transition Model) as well as how to send and receive text messages on their mobile phone. Following discharge to home, the virtual nurse will continue to coach Veterans and their family members and improve post-discharge access to care through two-way computer-tailored text messaging made possible by VHA's new HealtheDialog system. Specific aims are to:

1. Refine methods and collect formative measures to guide implementation
2. Conduct a randomized trial of the technology-assisted care transition intervention
3. Evaluate the intervention, including its effectiveness, implementation, and budget impact

The investigators propose a mixed methods formative assessment and simulation experiment to refine existing technologies to the VA care transition setting (Aim 1). This will be followed by a multi-site randomized type1 hybrid implementation trial (Aims 2 and 3). The trial will evaluate the effectiveness of the virtual nurse intervention in twelve clinical teams and also gather information about its implementation to inform broader rollout.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Diagnosis of chronic heart failure or chronic obstructive pulmonary disease
* Admission to a general medical service
* Able and willing to engage with touchscreen technology
* Have a text-enabled cellular phone to receive the post-discharge text messages

Exclusion Criteria:

* Not Veterans
* Not diagnosed of chronic heart failure or chronic obstructive pulmonary disease
* Not admitted to a general medical service
* Not capable of using touchscreen technology
* Do not have a text-enabled cellular phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Patrick Hogan, PhD MS BS, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (5):
- United States (5):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: In-patient virtual nurse on-screen touchscreen and outpatient virtual nurse follow-up by texting
Period: Overall Study
Arm/Group | Intervention | Active Attention Control
Started | 80 | 60
Completed | 57 | 50
Not Completed | 23 | 10
Not completed — Lost to Follow-up | 14 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Did not receive allocated protocol (did not enroll in texting program) | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Technology-assisted Care Transition Arm | Active Attention Control | Total
Number analyzed (Participants) | 80 | 60 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 43
  >=65 years | 55 | 42 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.01 (8.40) | 68.40 (7.70) | 68.705 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 78 | 59 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 77 | 58 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 66 | 42 | 108
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 60 | 140
Problems learning about medical conditions [Count of Participants; unit: Participants] — We administered a health literacy screening question, "How often do you have problems learning about your medical condition because of difficulty understanding written information?" We scored the responses on a five-point Likert scale (always; often; sometimes; occasionally; never) from 1 to 5, with a score range of 1-5, with a higher score indicating fewer problems learning about their medical conditions.
  Participants
    Always | 2 | 6 | 8
    Often | 3 | 1 | 4
    Sometimes | 2 | 9 | 11
    Occasionally | 14 | 5 | 19
    Never | 57 | 39 | 96
    No response | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pre-post Change in Combined Emergency and Urgent Care Service Utilization
Description: Comparing Total Number of Combined Emergency and Urgent Care Utilization for Veterans with CHF and/or COPD between Intervention and Control across time. This measure is defined as the total number of VA emergency department visits and VA urgent care visits for each participant during the study period.
Time Frame: 18 months prior to enrollment and 12 months post-discharge
Population: Enrolled Veterans who had complete data for this measure
Measure: Mean (Standard Deviation); unit: care utilization events
Groups:
- Intervention: Technology-assisted care transition intervention: In-patient virtual nurse on-screen touchscreen and outpatient virtual nurse follow-up by texting
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 79 | 59
care utilization events
  Pre-Trial Utilization | 1.06 (3.05) | 1.03 (2.67)
  Post-Trial Utilization | 0.92 (2.86) | 0.71 (1.78)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — Using a pre-intervention rate of 18 for both intervention and control, and a post-control change of 1, assuming an alpha of 0.05, we have power (0.8) to detect a difference of differences in change in mean urgent care/ED utilization of 0.75 with a standard deviation equal to the control mean; however, the equivalence boundary did not apply because this is a pragmatic trial; p = 0.45, Mixed Effects Negative Binomial Model; A segmented negative binomial regression model was used to estimate changes in ED/urgent care utilization between the intervention and control groups; Incidence Rate Ratio = 1.11, 95% CI 2-sided [0.85 to 1.45], Standard Error of Mean 0.15

2. Secondary Outcome: Care Transition Measure (CTM) Score Comparison
Description: The Care Transition Measure (CTM) is a validated, 15-item instrument used to measure the quality of a patient's care transition. The CTM has been shown to discriminate between patients discharged from the hospital who did and did not have a subsequent emergency department visit or rehospitalization for their index condition. Each of the CTM items has a 4-point Likert response scale ranging from 1 (strongly disagree) to 4 (strongly agree). When scoring the CTM, the lowest possible score is 0 and the highest possible score is 100, where higher scores indicate a better quality care transition.
Time Frame: Responses to the CTM were collected from the intervention and control groups 7 days post-discharge.
Population: Enrolled Veterans who had complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 80 | 59
score on a scale | 75.96 (13.90) | 77.00 (14.41)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — We initially powered at 80% to detect an effect size of 0.5 for all secondary outcomes; however, the equivalence boundary did not apply because this is a pragmatic trial; p = 0.05, Mixed Models Analysis; Beta for the Mean Difference = -1.80, 95% CI 2-sided [-7.21 to 3.61]

3. Secondary Outcome: Adherence to Refills and Medications Scale (ARMS) Score Comparison
Description: The Adherence to Refills and Medication Scale (ARMS) is a validated, 12-question instrument that assesses patient medication adherence across all literacy levels. Additionally, ARMS can be used to identify potential adherence barriers. The ARMS uses a 4-point Likert scale ranging from 1 (none of the time) to 4 (all of the time). The score range is 12-48 with lower scores indicating better adherence.
Time Frame: ARMS questionnaires were given to all participants at baseline and again at 30-day post-discharge follow-up
Population: Enrolled Veterans with CHF and/or COPD who completed baseline and 30-day follow-up and had complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 63 | 48
score on a scale
  Baseline Score | 15.24 (2.61) | 16.91 (5.03)
  30-Day Follow-Up Score | 15.0 (1.71) | 15.0 (2.26)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.03, Mixed Models Analysis; MMA by group, time, and group by time as predictors. We also adjusted by: Marital Status and indicator variable for problems learning online; Beta for the Mean Difference = 0.82, 95% CI 2-sided [0.08 to 1.57], Standard Error of Mean 0.38

4. Secondary Outcome: Health Distress Score Comparison
Description: We used the Lorig Health Distress Scale to assess overall health-related distress. This 4-item instrument uses a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time). The score range is 0-5 with a higher score indicating more distress about health.
Time Frame: The Health Distress measure was assessed at baseline, 7 days post-discharge, and 30 days post-discharge.
Population: Enrolled Veterans with CHF and/or COPD who completed baseline, 7-day, and 30-day follow-up and had complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline Score | 3.48 (1.33) | 3.27 (1.58)
  30-Day Follow-Up Score | 2.90 (1.34) | 2.79 (1.36)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.75, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Beta for Mean Difference = -0.06, 95% CI 2-sided [-0.41 to 0.29], Standard Error of Mean 0.18

5. Secondary Outcome: Self Efficacy for Managing Chronic Disease Scale Comparison
Description: The Self-Efficacy for Managing Chronic Disease Scale is a validated instrument that assesses symptom control, role, and emotional functioning. This 6-question instrument uses a 1-10-point scale ranging from 1 (not at all confident) to 10 (totally confident). The score range is 1-10 with higher scores indicating higher self-efficacy.
Time Frame: Baseline and 30-day follow-up.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline Score | 6.23 (2.32) | 6.29 (2.52)
  30-Day Follow-Up Score | 6.34 (2.13) | 6.21 (2.59)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.74, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Beta for Mean Difference = 0.10, 95% CI 2-sided [-0.50 to 0.70], Standard Error of Mean 0.30

6. Secondary Outcome: Outcome Measure Title: Self-Care of Heart Failure Index Score Comparison
Description: The Self-Care of Heart Failure Index, version 6.2, is a validated instrument that assesses patient management and maintenance of their heart failure and uses a 4-point Likert scale ranging from 1 (never or rarely) to 4 (always or daily). We used the maintenance subscale of this instrument which includes 10 items that measure daily activities known to assist in the health of heart failure patients. The score range is 10 to 100 with higher scores indicating better patient self-management.
Time Frame: Baseline and 30-day follow-up
Population: Enrolled Veterans with CHF who completed baseline and 30-day follow-up and had complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 45 | 38
score on a scale
  Baseline Score | 28.51 (5.62) | 27.20 (6.22)
  -Day Follow-Up Score | 31.11 (5.92) | 30.71 (5.63)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.63, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Beta for mean difference = -0.41, 95% CI 2-sided [-2.21 to 1.29], Standard Error of Mean 0.87

7. Secondary Outcome: COPD Self-Management Scale Score Comparison
Description: The COPD Self-Management Scale by Zhang is a validated instrument to assess patient self-management of COPD and uses a 5-point Likert scale ranging from 1 (never) to 5 (always). We used 10 question items from this instrument that measure common activities associated with the management of COPD. The scoring range is 10-50, with higher scores indicating better COPD self-management.
Time Frame: Baseline and 30-day follow-up
Population: Enrolled Veterans with COPD who completed baseline and 30-day follow-up and had complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 24 | 14
score on a scale
  Baseline Score | 37.91 (6.58) | 36.95 (6.29)
  30-Day Follow-Up Score | 39.58 (5.65) | 35.71 (4.86)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.23, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Beta of Mean Difference = 1.54, 95% CI 2-sided [-0.97 to 4.05], Standard Error of Mean 1.26

8. Secondary Outcome: Self-Efficacy for Managing Symptoms (PROMIS)
Description: The Self-Efficacy for Managing Symptoms scale is a 4-question, validated measure and is a part of the larger Patient-Reported Outcomes Measurement Information System (PROMIS) used to assess physical, mental, and social health in patients with chronic conditions. We used the 4-question items from this scale with response options on a 6-point Likert scale ranging from 1 (not at all confident) to 6 (very confident). The scoring range is 4-24, with higher scores indicating higher self-efficacy for symptom management.
Time Frame: Enrolled Veterans with CHF and/or COPD who completed baseline and 30-day follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline Score | 17.87 (5.28) | 18.20 (5.17)
  30-Day Follow-Up Score | 18.87 (4.64) | 17.53 (5.62)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.38, Mixed Models Analysis — MMA by group, time, and group by time as predictors. We also adjusted by: Marital Status and indicator variable for problems learning online; Beta for the Mean Difference = -2.43, 95% CI 2-sided [-7.95 to 3.10], Standard Error of Mean 2.80

9. Secondary Outcome: Self-Efficacy for Managing Medications and Treatments (PROMIS)
Description: The Self-Efficacy for Managing Medications and Treatments scale is a 4-question, validated measure and is a part of the larger Patient-Reported Outcomes Measurement Information System (PROMIS) used to assess physical, mental, and social health in patients with chronic conditions. We used the 4-question items from this scale with response options on a 6-point Likert scale ranging from 1 (not at all confident) to 6 (very confident). The scoring range is 4-24, with higher scores indicating higher self-efficacy for managing medications and treatments.
Time Frame: Enrolled Veterans with CHF and/or COPD who completed baseline and 30-day follow-up.
Population: Enrolled Veterans with CHF and/or COPD who completed baseline and 30-day follow-up and completed data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Active Attention Control
Number analyzed (Participants) | 63 | 49
score on a scale
  Baseline Score | 18.89 (5.42) | 18.63 (4.88)
  30-Day Follow-Up Score | 19.08 (4.54) | 18.12 (5.36)
Statistical Analysis 1: Comparison: Intervention vs Active Attention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.38, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Beta for the Mean Difference = -2.79, 95% CI 2-sided [-9.10 to 3.52], Standard Error of Mean 3.20

ADVERSE EVENTS:
Time Frame: Study participants were monitored for adverse events during the active enrollment period of thirty (30) days from their hospital discharge date.
Description: In monitoring, collecting, and reporting data, the study did not consider rehospitalization to be a serious adverse event as the primary outcome of focus was healthcare utilization, including rehospitalization. The target population for this study, hospitalized Veterans with congestive heart failure and/or chronic obstructive pulmonary disease, tends to be older, sicker, and faced with more complex medical needs. For these reasons, rehospitalization can be common among this population.
Arm/Group | Technology-assisted Care Transition Arm | Active Attention Control
All-Cause Mortality (participants affected / at risk) | 24/80 | 21/60
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/60
Other Adverse Events (participants affected / at risk) | 0/80 | 0/60

LIMITATIONS AND CAVEATS:
It is important to interpret the results in light of this study's sample size limitations. Enrollment was slow and compounded by a recruitment halt during COVID-19. While we believe that we have a sufficient sample to examine utilization outcomes, enrollment was still less than anticipated. Lastly, it can be difficult to determine meaningful differences for the secondary outcomes used in this study, especially in light of the complex patient population and the novelty of the intervention tested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT02632552/Prot_SAP_000.pdf
  • Informed Consent Form (2013-09-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT02632552/ICF_001.pdf